CLINICAL TRIAL: NCT07371715
Title: Efficacy, Safety, and Feasibility of a Home-Based Auricular Transcutaneous Electrical Stimulation Intervention Using a Low-Frequency TENS-Like Device to Improve Sleep Quality and Psycho-Academic Outcomes in Health Sciences Students: A Randomized Controlled Pilot Study
Brief Title: Home-Based Auricular Transcutaneous Vagus Nerve Stimulation (tVNS) for Sleep Quality and Psycho-Academic Outcomes in Health Sciences Students
Acronym: NEUROSLEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Ismael Romero García, Principal Investigator / PhD Candidate, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AURI-tVNS-SLEEP-2026; CEIH-UPO: 25/1-17 (Other: Ethics Committee Approval Code (CEIH, UPO))
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbances; Insomnia; Stress
Keywords: Transcutaneous Vagus Nerve Stimulation; sleep quality; Auricular Stimulation; university students
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, two-arm, parallel-group pilot trial (1:1 allocation).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to group allocation. Outcome assessors and data analysts are blinded to treatment assignment. The control condition consists of stimulation applied to the earlobe to mimic sensory stimulation without active auricular vagal stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Experimental): Home-based auricular transcutaneous vagus nerve stimulation (tVNS) applied to the left cymba conchae (or tragus if needed) using a low-frequency TENS-like device. Sessions are performed for 60 minutes, 5 days/week for 3 weeks. Stimulation intensity is adjusted to a strong but comfortable paresthesia below pain threshold.
  Interventions: Device: Auricular Transcutaneous Vagus Nerve Stimulation (tVNS)
- Control (Earlobe Stimulation) (Placebo Comparator): Control stimulation delivered to the ipsilateral earlobe using the same device and schedule as the active intervention (60 minutes, 5 days/week for 3 weeks) to mimic sensory stimulation without targeting auricular vagal afferents.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Auricular Transcutaneous Vagus Nerve Stimulation (tVNS) — Home-based auricular transcutaneous vagus nerve stimulation (tVNS) delivered using a low-frequency TENS-like device. Stimulation is applied to the left cymba conchae (or tragus if needed) for 60 minutes per session, 5 sessions per week for 3 weeks. Biphasic symmetrical waveform (25 Hz, 200 μs pulse width). Intensity is individually adjusted to a strong but comfortable paresthesia below pain threshold.
  Arms: Active tVNS
Device: Sham stimulation — Control stimulation delivered using the same low-frequency TENS-like device and parameters (25 Hz, 200 μs) applied to the ipsilateral earlobe to mimic sensory stimulation. Sessions are performed for 60 minutes per session, 5 sessions per week for 3 weeks, without targeting auricular vagal afferents.
  Arms: Control (Earlobe Stimulation)

SUMMARY:
This study aims to evaluate the efficacy, safety, and feasibility of a home-based auricular transcutaneous vagus nerve stimulation (tVNS) program in Health Sciences university students with poor sleep quality. Participants will be randomly assigned (1:1) to receive either active auricular stimulation (cymba conchae/tragus) or a control stimulation applied to the earlobe. The intervention will be self-administered at home using a low-frequency TENS-like device for 60 minutes per session, 5 sessions per week for 3 weeks. Sleep quality will be primarily assessed using the Pittsburgh Sleep Quality Index (PSQI) before and after the intervention. Secondary outcomes include insomnia severity, daytime sleepiness, perceived stress, anxiety, quality of life, and psycho-academic outcomes.

DETAILED DESCRIPTION:
Sleep disturbances are highly prevalent among university students and are frequently associated with academic stress and impaired psycho-academic functioning. Transcutaneous vagus nerve stimulation (tVNS) is a non-invasive neuromodulation approach with potential to modulate autonomic function and stress responses, which may contribute to improvements in sleep quality.

This study is designed as a randomized controlled pilot trial to assess the efficacy, safety, and feasibility of a home-based auricular tVNS intervention in Health Sciences university students. Eligible participants will be aged 18-35 years and will present poor sleep quality (PSQI > 7) and primary insomnia criteria. Participants will be recruited from two academic centers (University of Malaga and Centro Universitario San Isidoro, affiliated with Pablo de Olavide University, Seville) and will be randomly allocated (1:1) to one of two arms: (1) active auricular stimulation targeting the left cymba conchae (with tragus as an alternative if needed), or (2) control (sham) stimulation delivered to the ipsilateral earlobe. Randomization will be performed using block randomization, and outcome assessors and data analysts will remain blinded to group assignment.

The intervention will be delivered at home using a low-frequency TENS-like device with biphasic symmetrical waveform (25 Hz, 200 μs pulse width), administered for 60 minutes per session, 5 sessions per week for 3 weeks. Stimulation intensity will be individually adjusted to achieve a clear but comfortable paresthetic sensation below the pain threshold. Adherence will be monitored using an electronic diary with time stamps and daily photographic verification of electrode placement.

The primary outcome is sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI) pre- and post-intervention. Secondary outcomes include insomnia severity (ISI), daytime sleepiness (ESS), perceived stress (PSS-14), anxiety measures (e.g., BAI and HAMA), depressive symptoms (HAMD), fatigue (FFS), and health-related quality of life (SF-12 v2). Psycho-academic outcomes will be measured using self-reported GPA and credits passed at the end of the semester. Safety will be assessed through systematic recording of adverse events throughout the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35 years.
* Undergraduate student enrolled in a Health Sciences degree program.
* Poor sleep quality defined as PSQI > 7.
* Meets diagnostic criteria for primary insomnia according to ICSD-3.
* Ability to understand study procedures and provide written informed consent.
* Willing and able to self-administer the intervention at home and complete study questionnaires.

Exclusion Criteria:

* Current severe psychiatric disorder or ongoing psychotherapy treatment.
* Neurological disorders (e.g., epilepsy).
* Cardiac arrhythmias or implanted cardiac devices (e.g., pacemaker).
* Current use of medications that significantly affect sleep (e.g., hypnotics or anxiolytics), unless stable and approved by the investigator.
* Pregnancy.
* Ear infection, skin lesions, or dermatologic condition preventing electrode placement.
* Hypersensitivity or intolerance to electrical stimulation.
* Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline and end of week 3
  PSQI total score (0-21). Higher scores indicate worse sleep quality.
Anxiety Symptoms (Beck Anxiety Inventory, BAI) | Baseline and end of week 3
  BAI total score. Higher scores indicate greater anxiety symptoms.

SECONDARY OUTCOMES:
Insomnia Severity (Insomnia Severity Index, ISI) | Baseline and end of week 3
  ISI total score. Higher scores indicate greater insomnia severity.
Daytime Sleepiness (Epworth Sleepiness Scale, ESS) | Baseline and end of week 3
  ESS total score. Higher scores indicate greater daytime sleepiness.
Perceived Stress (Perceived Stress Scale-14, PSS-14) | Baseline and end of week 3
  PSS-14 total score. Higher scores indicate greater perceived stress.
Quality of Life (12-Item Short Form Survey, SF-12 v2) | Baseline and end of week 3
  SF-12 v2 component summary scores (physical and mental). Higher scores indicate better health-related quality of life.
Academic Performance (GPA and Credits Passed) | Baseline and end of semester (up to 16 weeks)
  Self-reported grade point average (GPA) and number of credits passed during the academic term.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to data protection regulations and participant privacy requirements. Study results will be reported in aggregate form. De-identified data may be made available upon reasonable request and with approval from the investigators and the ethics committee, in accordance with applicable regulations.